CLINICAL TRIAL: NCT00134667
Title: A Phase IIIb/IV Randomized, Double-Masked, Active Controlled, Dose-Ranging, Multi-Center Comparative Trial, in Parallel Groups, to Compare the Safety and Efficacy of Intravitreal Injections of Pegaptanib Sodium (Macugen) Given Every 6 Weeks for 102 Weeks, to Pegaptanib Sodium Plus Photodynamic Therapy (PDT) With Visudyne, in Patients With Exudative Age-Related Macular Degeneration (AMD)
Brief Title: Macugen (Pegaptanib Sodium) Alone, Versus Macugen in Combination With PDT (Photodynamic Therapy) With Visudyne (Verteporfin) in Patients With Age-Related Macular Degeneration (AMD)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Eyetech Pharmaceuticals (Industry)
Collaborators: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EOP1012
Record Dates: First submitted 2005-08-24; First posted 2005-08-25 (Estimated); Last update posted 2007-01-15 (Estimated); Status verified 2007-01

CONDITIONS: Age-Related Macular Degeneration
Keywords: AMD; Age-Related Macular Degeneration; Macular Degeneration; Macugen; Photodynamic Therapy; PDT; Visudyne; pegaptanib sodium; verteporfin; Predominantly Classic; Age-Related Macular Degeneration (AMD)
MeSH Terms: conditions — Macular Degeneration | interventions — Photochemotherapy; 1-phenyl-3,3-dimethyltriazene; Verteporfin; pegaptanib

INTERVENTIONS:
Drug: Photodynamic Therapy (PDT) with Visudyne (verteporfin)
Drug: Macugen (pegaptanib sodium)

SUMMARY:
The purpose of the trial is to compare whether Macugen (pegaptanib sodium) in combination with PDT with Visudyne (verteporfin) is safe and effective in slowing down the leakage of fluid within the eye and thereby stabilizing or improving vision when compared to Macugen alone. Patients must be recently diagnosed with predominantly classic wet AMD and must be eligible for PDT.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of either gender; aged 50 years or greater.
* Subfoveal choroidal neovascularization (CNV) due to AMD with predominantly classic lesion composition
* Best corrected visual acuity in the study eye between 20/40 and 20/200

Exclusion Criteria:

* Any prior PDT with Visudyne to the study eye
* Any previous AMD thermal laser therapy to the study eye

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360
Dates: Start 2005-03; Study Completion 2008-10

CONTACTS AND LOCATIONS:
Locations (1):
- Retina Centers, P.C., Northwest Location, Tucson, Arizona, United States